CLINICAL TRIAL: NCT06053840
Title: An Open-label Trial to Evaluate the Safety and Efficacy of Chloral Hydrate in Patients with Severe Insomnia
Acronym: RESTORE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmanovia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1007757
Record Dates: First submitted 2023-06-21; First posted 2023-09-26 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Insomnia; Insomnia Chronic; Chloral Hydrate
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Chloral Hydrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Chloral Hydrate

INTERVENTIONS:
Drug: Chloral Hydrate — Participants will be involved in the trial for approximately 7-8 weeks, the first week to collect baseline data and complete screening and eligibility confirmation, the following two weeks they will administer IMP, and there will be a further 4 week observation period. All trial recruitment and follow-up procedures will be conducted remotely via telephone/video calls.

SUMMARY:
The primary aim of this Real-World Evidence trial is to establish whether short-term (2 weeks) treatment of Chloral Hydrate is effective in patients with severe insomnia which is interfering with normal daily life, and where other behavioural and pharmacologic therapies have failed in a real world setting.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years and ≤75 years
* Participant is willing and able to give informed consent
* Clinically significant impairment from severe insomnia (eg. ISI score 22-28)
* Previous treatment with sleep therapies (behavioural and pharmacologic), which have failed. Defined as the presence of ongoing severe insomnia (ISI score 22-28), despite previous use of other sleep therapies.
* Able to adhere to trial procedures
* Willingness to take a pregnancy test prior to starting IMP treatment (participants of childbearing potential)

Exclusion Criteria:

* Pregnant or breastfeeding
* Taking any substances that significantly affect sleep during the 2 week IMP treatment period
* Starting any new behavioural sleep therapies* during the 2 week IMP treatment period
* At point of enrolment taking substances that affects sleep at greater than maximum licensed doses
* Other sleep diagnosed/suspected sleep disorders (restless legs, periodic limb movements, unusual sleep timings (indicative of advanced/delayed sleep, etc), parasomnias
* Known severe hepatic impairment
* Known moderate / severe renal impairment / eGFR <60
* Known severe sleep apnea
* Known severe cardiac disease
* Known cardiac disease with QT prolongation
* History of myocardial infarction in the last 12 months
* History of stroke or TIA
* Taking medication that may cause QT prolongation
* Active gastritis, oesophagitis, gastric or duodenal ulcers or perforation
* Susceptible to acute attacks of porphyria
* Hypersensitivity to Chloral Hydrate or to any of the excipients (glycerol, liquid glucose, citric acid, sodium citrate, sodium benzoate, saccharin sodium, essence of passion fruit [containing natural flavouring, artificial flavouring, propylene glycol], and purified water)
* Individuals with a history of alcohol or drug abuse or dependence
* Patients taking antipsychotic medication in last 12 months
* History of overdose or attempted overdose
* History of significant psychiatric disease
* Patients are taking one of the drugs listed as interacting with Chloral Hydrate and would need to continue taking these during the trial: alcohol, CNS depressants, antipsychotics, hypnotics, anxiolytics/sedatives, antidepressant agents, centrally acting muscle relaxants, narcotic, analgesics, anti-epileptic drugs, anaesthetics and sedative antihistamines, intravenous furosemide, anticoagulants.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational product in the past 4 months
* Participants of childbearing potential (participants who are anatomically and physiologically capable of becoming pregnant), or have a partner of childbearing potential, not willing to use highly effective contraceptives** for the duration of the trial, and who do not confirm a negative pregnancy test prior to starting the IMP.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
To assess the effectiveness of Chloral Hydrate in reducing insomnia severity | Self-rated insomnia severity, assessed at baseline and 2 weeks
  Change in self-rated insomnia severity, assessed using the Insomnia Severity Index

SECONDARY OUTCOMES:
To explore whether Chloral Hydrate will affect Self-rated insomnia severity, assessed at baseline and 2 weeks | Self-rated insomnia severity, assessed at baseline, 1 week and 6 weeks
  Change in self-rated insomnia severity, assessed using the Insomnia Severity Index (ISI)
To explore whether Chloral Hydrate will affect Daytime sleepiness | Epworth Sleepiness Scale scores, assessed at baseline, 1 week, 2 weeks and 6 weeks
  Change in Epworth Sleepiness Scale scores which is based on a 0-3 scale with 0 being No chance of dozing, and 3 High chance of dozing.
To explore whether Chloral Hydrate will affect Insomnia severity | Self-rated insomnia severity, assessed at baseline, 1 week and 6 weeks
  Change in self-rated insomnia severity, assessed using the Insomnia Severity Index (ISI)
To explore whether Chloral Hydrate will affect Health-related quality of life | SF-36 and EQ-5D-5L responses, assessed at baseline, 1 week, 2 weeks and 6 weeks
  Change in health-related quality of life, measured using the ShortForm 36 (SF-36) and EQ-5D-5L questionnaires. The SF-36 is based on a 1-5 with 1 being excellent and 5 poor. EQ-5D-5L is scored on a 0-100 scale with 0being the worst health possible, and 100 the best health you can imagine.
To explore whether Chloral Hydrate will affect anxiety and Depression | HADS scores, assessed at baseline, 1 week, 2 weeks and 6 weeks
  Change in Hospital Anxiety and Depression Scale (HADS) scores. The scale is based on a 0-21 scale with 0-7 = Normal, 8-10 = Borderline abnormal (borderline case), 11-21 = Abnormal (case)
To explore whether Chloral Hydrate will affect Quality of sleep and sleep disturbances | PSQI responses assessed at baseline, 2 weeks and 6 weeks
  Change in Pittsburgh Sleep Quality Index (PSQI) scores
To investigate the safety of Chloral Hydrate | AEs and SAEs for the 6 week trial duration
  Evaluation of overall safety of Chloral Hydrate by the monitoring of AEs and SAEs
To investigate intervention adherence | Daily intervention adherence survey questions on days 1-14
  Daily intervention adherence for the duration of the intervention (2 weeks)
To assess tolerance of Chloral Hydrate | Total number of participants withdrawn from the IMP due to an AR
  Number of participants withdrawn from the IMP due to an AR, during the 2 week treatment period
To determine any reductions in the use of non-pharmacological sleep therapies | Non-pharmacological sleep therapies assessed at baseline, 1 week, 2 weeks and 6 weeks
  Change in use of non-pharmacological sleep therapies
To determine any reductions in 1. Concomitant prescribed medication 2. Over the counter medication used to facilitate sleep | 1. Concomitant medication assessed at baseline, 1 week, 2 weeks and 6 weeks 2. Over the counter medication used to facilitate sleep assessed at baseline, 1 week, 2 weeks and 6 week
  Change in
  1. Concomitant medication
  2. Over the counter medication used to facilitate sleep
Medical doctor assessment of effectiveness of Chloral Hydrate | CGI-S assessed at baseline, and CGI-I assessed at 2 weeks and 6 weeks
  Clinical Global Impressions - Severity Scale (CGI-S) assessed at baseline, and Clinical Global Impressions - Improvement scale (CGI-I) assessed after IMP treatment by the medically qualified doctor. Rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.

OTHER OUTCOMES:
To assess days off work | Percentage of days off work one month and 12 months prior to baseline, and assessed at 2 weeks (for the 2 week treatment period) and 6 weeks (for the 4 week observation period)
  Change in percentage of days off work

CONTACTS AND LOCATIONS:
Locations (1):
- Lindus Health, The Leather Market Weston Street, Bermondsey,, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No